CLINICAL TRIAL: NCT01663805
Title: Effects of the Use of "de Novo" Everolimus for the Expression of Cytokines in Kidneys From Extended Criteria Donors and With Delayed Graft Function
Brief Title: Effects of the Use of "de Novo" Everolimus in Renal Tranplant Population
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MARIO ABBUD FILHO (Other)
Responsible Party: Sponsor-Investigator, MARIO ABBUD FILHO, Principal Investigator, Instituto de Urologia e Nefrologia
Organization: Instituto de Urologia e Nefrologia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001ABR21T
Record Dates: First submitted 2012-04-12; First posted 2012-08-13 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-04

CONDITIONS: Delayed Function of Renal Transplant
Keywords: Extended Criteria Donor; Delayed Graft Function; DGF; Deceased donors aged ≥ 60 years; aged between 50 and 59 years; history of systemic hypertension; terminal creatinine levels > 1.5 mg/dL; death by a cerebrovascular accident
MeSH Terms: conditions — Delayed Graft Function | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everolimus (Active Comparator): SCD/ECD: BXB (2x20mg, D1 and D4) + EVL (3.0 -8.0ng/ml) + MYF (1440mg/d)+ Prednisone
  Interventions: Drug: Everolimus
- mycophenolate sodium (No Intervention): SCD/ECD: BXB (2x20mg, D1 and D4) + TAC + MYF (1440mg/d)+ Prednisone

INTERVENTIONS:
Drug: Everolimus — Everolimus is started immediately after transplantation, the dosage of 1.5 mg twice a day, adjusted to achieve and maintain the blood level of 3-8 ng/mL.
  Other Names: Certican
  Arms: Everolimus

SUMMARY:
This is an open, randomized, single-center study. The selected patients will be first divided into two major groups according to the type of organ to be transplanted: standard criteria donor (SCD) or extended criteria (ECD) kidney. Then, each group will be randomly allocated to one of the treatments: tacrolimus (TAC) or everolimus (EVL).

All patients received induction therapy with basiliximab (BXB) and maintenance with Mycophenolate Sodium (MYF) and prednisone (P). This study will evaluate as Primary objectives: To characterize the molecular profile of cytokines in kidneys obtained from deceased donors such as "standard" (SCD) and extended criteria (ECD) in biopsies taken before and after transplantation and to evaluate the effect of treatment with everolimus (EVL) in the expression of these molecules. And as Secondaries objectives: To correlate the pattern of cytokines with delayed graft function (DGF), cold ischemia time, episodes of acute rejection and patient and graft survival.

DETAILED DESCRIPTION:
A total of 80 patients will participate in the study, being distributed into 4 groups of 20 individuals. In a pilot study to assess the interventional effect of the mmediate use of EVL on the cytokine profile of ECD and SCD kidneys, compared to conventional immunosuppressive therapy with TAC, no statistical power analysis could be performed a priori.

Definitions of Extended Criteria Donor and Delayed Graft Function (DGF) Deceased donors aged ≥ 60 years or aged between 50 and 59 years and with at least two of the following risk factors: history of systemic hypertension terminal creatinine levels > 1.5 mg/dL or death by a cerebrovascular accident.

DGF (delayed graft function) is defined as the need for dialysis in the first 7 days after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (black and white subjects);
* End-stage renal disease with indication for transplantation (primary deceased-donor kidney transplant)
* "Standard" traditional (SCD) or extended criteria (ECD) donor;
* Informed consent form duly signed before SCD or ECD kidney transplantation.

Exclusion criteria:

* The subject, in the opinion of the investigator, is not able to complete the study protocol;
* Recipient of live-donor kidney graft;
* Multiple organ transplant recipient;
* Evidence of large systemic or localized infection;
* Evidence of infiltration, cavitation or consolidation on chest X-rays obtained during the evaluation in the screening / baseline visit;
* Use of any drug under investigation or treatment until up to 4 weeks before transplantation;
* Known or suspected hypersensitivity to tacrolimus, everolimus or mycophenolate sodium;
* Immunosuppressive therapies in addition to those described for this study;
* Hypersensitized patients (PRA > 30%);
* Patients with HIV+ or Hepatitis B or C virus infection.
* Patients for whom T0 and T15 biopsies were not taken.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Molecular profile of cytokines | 12 months
  To characterize the molecular profile of cytokines in kidneys obtained from deceased donors such as "standard" (SCD) and extended criteria (ECD) in biopsies taken before and after transplantation and to evaluate the effect of treatment with everolimus (EVL) in the expression of these molecules.

SECONDARY OUTCOMES:
Pattern of cytokines with DGF, cold ischemia time, episodes of acute rejection | 12 months
  To correlate the pattern of cytokines with DGF, cold ischemia time, episodes of acute rejection and patient and graft survival

CONTACTS AND LOCATIONS:
Overall Officials: Mario Abbud, MD.PhD, Principal Investigator — Instituto de Urologia e Nefrologia
Locations (1):
- Instituto de Urologia e Nefrologia, São José do Rio Preto, São Paulo, Brazil